CLINICAL TRIAL: NCT00335075
Title: A Multicenter, Open-Label, Randomized, Active-Controlled Parallel Groups Study Comparing the Efficacy and Safety of Temodal vs Semustine in the Treatment of Subjects With Recurrent Glioblastoma or Anaplastic Astrocytoma
Brief Title: Efficacy and Safety of Temodal vs Semustine in Subjects With Recurrent Glioblastoma or Anaplastic Astrocytoma (Study P03644)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03644
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Glioblastoma; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Temozolomide; Semustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temodal group (Experimental): Subjects treated with temozolomide.
  Interventions: Drug: Temozolomide
- Semustine group (Active Comparator): Subjects treated with semustine.
  Interventions: Drug: Semustine

INTERVENTIONS:
Drug: Temozolomide — Temozolomide orally for 5 consecutive days (Day 1 through Day 5) every 28 days, at a dose of 150 mg/m2/day for subjects previously treated with chemotherapy, or 200 mg/m2/day for subjects who have not received previous chemotherapy.
  Other Names: Temodal; Temodar; SCH 052365
  Arms: Temodal group
Drug: Semustine — Semustine orally once every 28 days at a dose of 150 mg/m2/day.
  Other Names: Methyl-CCNU
  Arms: Semustine group

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of temozolomide compared to semustine in the treatment of patients with glioblastoma multiforme or anaplastic astrocytoma.

ELIGIBILITY:
Inclusion Criteria:

* Prior histologic confirmation of glioblastoma, anaplastic astrocytoma.
* Evidence of tumor progression or recurrence.
* Age >=18 years.
* Karnofsky performance status >=60%.
* Absolute neutrophil count >=1,500/mm^3, platelet count >=100,000/mm^3, hemoglobin >=8g/dL.
* Serum BUN and creatinine <1.5 times upper normal limit of testing laboratory (ULN).
* Total bilirubin and direct bilirubin <1.5 times ULN.
* SGOT, SGPT <3 times ULN; alkaline phosphatase <2 times ULN.
* Life expectancy greater than 3 months.
* Informed consent obtained.
* If palliative radiation is needed, agree to give it prior to initiating chemotherapy with study drug. If palliative radiation is required during treatment with study drug, the patient should be permanently discontinued from further treatment with study drug.
* Women of childbearing potential must use a medically accepted, effective method of contraception.
* Women of childbearing potential must have a negative serum pregnancy test 24 hours prior to administration of study drug.

Exclusion Criteria:

* Chemotherapy (excluding nitrosourea, mitomycin C or vincristine), biologic therapy or immunotherapy within 4 weeks, inclusive, prior to study drug administration.
* Nitrosourea or mitomycin C administration within 6 weeks, inclusive, prior to study drug administration.
* Vincristine within 2 weeks prior to study drug administration.
* Completion of radiation therapy, interstitial brachytherapy or radiosurgery within 4 weeks prior to study drug administration.
* Surgery within 3 weeks, inclusive, prior to study drug administration.
* Acute infection requiring intravenous antibiotics.
* Frequent vomiting or medical condition that could interfere with oral medication intake (eg, partial bowel obstruction).
* Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
* Known HIV positive or AIDS-related illness.
* Pregnant or nursing women.
* Men who are not advised to use an effective method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-03-02 (Actual); Primary Completion 2006-02-23 (Actual); Study Completion 2006-02-23 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 months, 3 months, and 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months
Objective response | 6 months
Scoring of health-related quality of life | 6 months

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html